CLINICAL TRIAL: NCT07369973
Title: Respiratory Biofeedback Added to Strengthening Training in Patients With Chronic Kidney Disease
Acronym: RESPI-REN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SICEIA-2024-003384
Record Dates: First submitted 2026-01-08; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (Stages 4 and 5)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Participants will receive diaphragmatic biofeedback combined with respiratory muscle training three times per day for 6 weeks
  Interventions: Other: Diaphragmatic biofeedback combined with respiratory muscle training
- Control Arm (Placebo Comparator): Placebo intervention based on conscious breathing three times per day for 6 weeks
  Interventions: Other: PLACEBO INTERVENTION

INTERVENTIONS:
Other: Diaphragmatic biofeedback combined with respiratory muscle training — This intervention is novel because it integrates diaphragmatic biofeedback into a structured respiratory muscle training program specifically designed for patients with chronic kidney disease, a population in which respiratory dysfunction is prevalent yet under-addressed. By providing real-time feedback on diaphragmatic activity, the intervention aims to enhance motor learning, improve activation of the diaphragm, and optimize training efficiency beyond conventional breathing or respiratory muscle training approaches.
  Arms: Treatment Arm
Other: PLACEBO INTERVENTION — The placebo intervention will consist of concious guided breathing sessions based on the participant's subjective respiratory sensations, without the use of objective physiological feedback or diaphragm-specific biofeedback. Participants will be instructed to follow standardized breathing guidance focused on perceived comfort and awareness, matching the intervention group in session frequency and duration.
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is to learn whether diaphragmatic biofeedback added to respiratory muscle training improves clinical and functional outcomes in adults with chronic kidney disease. It will also evaluate the feasibility and acceptability of this intervention.

The main questions it aims to answer are:

Is diaphragmatic biofeedback added to respiratory muscle training acceptable and well tolerated in patients with chronic kidney disease? Does this intervention reduce respiratory symptoms and complications in this population? Does diaphragmatic biofeedback added to respiratory muscle training improve cardiorespiratory capacity and quality of life? Researchers will evaluate diaphragmatic biofeedback combined with respiratory muscle training and a placebo intervention based on conscious breathing to assess its effects.

Participants will:

* Perform the assigned intervention three times per day for 6 weeks
* Follow a structured respiratory muscle training program with diaphragmatic biofeedback
* Be monitored for symptoms, respiratory complications, and perceived quality of life throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Diagnosis of chronic kidney disease (CKD) at any stage
* Clinically stable condition, with no acute medical events in the previous 4 weeks
* Ability to understand and follow breathing and training instructions
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Acute respiratory infection or unstable pulmonary disease
* Severe cognitive impairment or neurological condition limiting cooperation
* Unstable cardiovascular disease or contraindications to respiratory muscle training
* Recent thoracic or abdominal surgery (<3 months)
* Significant visual impairment that prevents proper use of the biofeedback device
* Participation in another interventional clinical trial during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events during intervention sessions | Baseline to 6 weeks
  Adverse events and discomfort related to the intervention will also be recorded to evaluate overall number of adverse events registered during intervention period.
Respiratory Symptoms assessed by Edmonton Symptom Assessment Scale (ESAS) | Baseline to 6 weeks
  Respiratory symptoms will be assessed using the validated symptom questionnaire and clinical reporting, focusing on perceived dyspnea and fatigue , and other respiratory-related complaints during daily activities. The Edmonton Symptom Assessment Scale (ESAS) is a validated instrument that assesses symptom severity, with each symptom rated on a numeric scale ranging from 0 (no symptom) to 10 (worst possible severity). Thus, higher scores indicate a worse outcome and greater symptom burden.
Respiratory Complications | Baseline to 12 weeks
  The occurrence of respiratory complications during the intervention period will be monitored and recorded, including any clinically relevant respiratory events reported by participants or identified during follow-up assessments.
Quality of Life of participants evaluated by Euqol-5Dimensions questionnaire | Baseline to 6 weeks
  Health-related quality of life will be assessed using a validated questionnaire to evaluate perceived physical, emotional, and functional well-being in participants undergoing the intervention. The EuroQol 5-Dimension (EQ-5D) questionnaire is a standardized measure of health-related quality of life comprising five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Health states are converted into a utility index score, typically ranging from values below 0 (worse than death) to 1 (full health), where higher scores indicate better health status; additionally, the EQ-5D includes a visual analogue scale (EQ-VAS) from 0 to 100, with higher scores reflecting better perceived health.
Acceptability of intervention considering number of sessions completed by participant | 6 weeks
  Acceptability of diaphragmatic biofeedback added to respiratory muscle training will be assessed through participant completion rates.

SECONDARY OUTCOMES:
Cardiorespiratory Capacity evaluated using 6 Minutes Walking test | Baseline to 6 weeks
  Changes in cardiorespiratory capacity will be evaluated using standardized functional or physiological assessments appropriate for patients with chronic kidney disease, aiming to determine whether the intervention improves respiratory and exercise-related capacity. The Six-Minute Walk Test (6MWT) measures functional exercise capacity by recording the total distance walked in six minutes, expressed in meters, with higher distances indicating better functional performance. There is no fixed minimum or maximum value, as results depend on the individual's physical capacity and clinical condition.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Heredia-Ciuró, PhD, Principal Investigator — Universidad de Granada; Marie Carmen Valenza, PhD, Study Director — Universidad de Granada

IPD SHARING:
Plan to Share IPD: Undecided